CLINICAL TRIAL: NCT04497506
Title: Wise Interventions for Adolescents and Young People in the Digital Society
Brief Title: Wise Interventions in the Digital Society
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Collaborators: Fundación BBVA (Unknown)
Responsible Party: Principal Investigator, Esther Calvete, Principal Investigator, Deusto Stress Research Team, University of Deusto, University of Deusto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR[18]_SOC_0096
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Cyberbullying; Grooming; Risk Behavior
Keywords: Adolescence; Youth; Cyberbullying; Grooming; Sexting; Prevention
MeSH Terms: conditions — Cyberbullying; Grooming; Risk-Taking

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio blocked by gender to one of two groups: experimental condition (SA+ITP) versus control condition (anti-stress condition) in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation will be concealed to the participants, researchers -who will be in class the assessment days if possible depending on the Covid-19 scenario- and teachers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-affirmation and Incremental theory of personality (Experimental): 1 hour Wise intervention (based on SA and ITP) consisting on several tasks to be completed online individually.
  Interventions: Behavioral: Wise Intervention (Self-affirmation and Incremental theory of personality)
- Standard preventive intervention (Other): 1 hour educational intervention (about stress management) consisting on several tasks to be completed online individually.
  Interventions: Behavioral: Standard preventive intervention

INTERVENTIONS:
Behavioral: Wise Intervention (Self-affirmation and Incremental theory of personality) — The intervention designed to promote prosocial behavior and reduce online risks is based on four general types of change strategies: (1) scientific knowledge, (2) generation of new meanings, (3) commitment through action, and (4) active reflection. It includes two components: a self-affirmation activity and an ITP intervention. The SA component includes a list of values so that they could choose the two or three most important for them. Next, they are asked to write why those selected values are the most important to them. The ITP component includes activities such as reading scientific information about social behavior and its role in people's well-being, the meaning and value of online risk behaviors through stories and videos of the experiences of other young people of their age, and self-persuasion exercises that involve an active commitment to change.
  Arms: Self-affirmation and Incremental theory of personality
Behavioral: Standard preventive intervention — It consists of an educational intervention that provides a number of strategies to manage everyday conflicts among adolescents. This intervention teaches them new ways to manage these difficulties through different actions (relaxation, distraction, sports, etc.). Finally, they are asked to plan the strategies they will use in the future in the face of some difficulties and to recommend some guidelines for another adolescent who may be going through a similar situation.
  Arms: Standard preventive intervention

SUMMARY:
This study evaluates the effectiveness of a Wise intervention based on self-affirmation (SA) and Implicit Theories of Personality (ITP) in Spanish adolescents and young people. Half of participants will receive the ITP and self-affirmation intervention, while the other half will receive a control intervention.

DETAILED DESCRIPTION:
Adolescence is a period that involves important transitions and learning opportunities. Adolescents and young people learn and develop new competencies and facets in the digital society. Hence, a large part of their social relationships takes place through social media.This offers them numerous positive opportunities for the emotional and social development of adolescents and young people. They can develop positive interactions through prosocial behaviors, empathy, and social support towards others. At the same time it is not without potential risks, especially in adolescence, a stage of psychological vulnerability for risky behaviors. Very recently, interest in scientific social psychology has grown due to a new approach to interventions, which have been called "wise interventions." This approach involves a set of rigorous techniques, based on theory and research, that address specific psychological processes to help people thrive in various life environments. The main objective of this project is to design and evaluate the effectiveness of a wise intervention based on self-affirmation (SA) and Implicit Theories of Personality (ITP) to promote various online prosocial behaviors (help, empathy, collaboration) and prevent online risk and harassment behaviors (online bullying, sexting, grooming). Secondary objectives are (1) to assess the moderating role of gender and the degree of evolutionary development of adolescents and young people, and (2) to evaluate potential mediating mechanisms for the effectiveness of the interventions. The study will involve the evaluation of the intervention in a sample of around 1000 young and adolescents randomly allocated to experimental and control condition.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the adolescents and their parents.
* To be fluent in Spanish and/or Euskera.

Exclusion Criteria:

* Lack of permission by parents and the adolescent.
* Lack of understanding of the instructions.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1212 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores of the Cyber Bullying Questionnaire (CBQ; Calvete et al., 2010; Gámez-Guadix, Villa-George, & Calvete, 2014) | Baseline, 3 months, and 6 months.
  Self reported levels of perpetration (9 items) and victimization (9 items) of peer cyber aggression. Each item is scored 0-4 (0 = never; 4 = almost every week).
Change from baseline scores of the Online Sexual Solicitation and Interaction of Minors with Adults Questionnaire (Gámez-Guadix, De Santisteban, & Alcazar, 2017). | Baseline, 3 months, and 6 months.
  Self reported items that assess the sexual interactions with an adult (10 items). Items are rated on a four-point response scale ranging from 0 (never) to 3 (6 or more times).
Change from baseline scores of the Sexting questionnaire (Gámez-Guadix, Almendros, Borrajo, & Calvete, 2015). | Baseline, 3 months, and 6 months.
  Self reported items about sending photos, information or videos of sexual or intimate content to three potential recipients: a partner, a friend and someone they have met on Internet but not in person (3 items). A five-point response scale was used ranging from 0 (never) to 4 (7 or more times).

SECONDARY OUTCOMES:
Change from baseline scores of the Online Prosocial Behavior Scale (OPBS; Erreygers, Vandebosch, Vranjes, Baillien y De Witte, 2017). | Baseline, 3 months, and 6 months.
  Self reported items about online prosocial behaviors (4 items). A five-point response scale was used ranging from 1 (never) to 5 (every day).
Change from baseline scores of the Cyber Dating Abuse Questionnaire (CDAQ; Borrajo et al., 2015) | Baseline, 3 months, and 6 months (only in participants with a dating relationship).
  Self reported items about dating aggressive behaviors of perpetration (4 items) and victimization (4 items). Items scored 0-3 (0 = never; 3 = almost always).
Change from baseline scores of the reduced version of the Center for Epidemiological Studies Depression (CES-D; Rueda-Jaimes et al., 2009). | Baseline, 3 months, and 6 months.
  Self reported symptoms of depression through 10 items, with a four-point response scale ranging from 0 (practically never) to 3 (almost all the time).

OTHER OUTCOMES:
Change from baseline scores of attitude towards cyberbullying measure | Baseline, intervention day, 3 months, and 6 months.
  Self reported ad hoc measures developed by the research team of the attitude towards cyberbullying. The participants will classify one situation of cyberbullying through adjectives using the semantic differential technique with a response range of 7 points.
Change from baseline scores of attitude towards different courses of action measure | Baseline, intervention day, 3 months, and 6 months.
  Self reported ad hoc measures developed by the research team of the attitude towards different courses of action when the adolescent witnesses cyberbullying. The participants will rate four different ways to react to cyberbullying through semantic differential items.
Change from baseline scores of the anticipation of reactions and behaviors measure | Baseline, intervention day, 3 months, and 6 months.
  Self reported ad hoc measures developed by the research team of the anticipation of reactions and behaviors when the adolescent is a witness. The participants will answer seven items on a five-point response scale ranging from 0 (totally disagree) to 3 (totally agree).
Change from baseline scores of Entity and incremental theories (Levy, Stroessner, & Dweck, 1998). | Baseline, intervention day, 3 months, and 6 months.
  Entity and incremental theories will be evaluated using eight items adapted to the situations of bullying in schools. Items are rated on a six-point scale ranging from 1 (strongly disagree) to 6 (strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Esther Calvete, PhD, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available at OSF when the results of the study are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol and informed consent protocol will be published at clinicaltrials.org Data will be available at OSF when the results are published.
Access Criteria: Public

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT04497506/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT04497506/ICF_001.pdf